CLINICAL TRIAL: NCT04041869
Title: Residential MapTrek- Increasing Physical Activity Among Older Adults in a Residential-Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Lucas Carr, Associate Professor, Department of Health & Human Physiology, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201904816; UL1TR002537 (NIH)
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Sedentary Behavior
Keywords: Older adults; Walking; Fitbit
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MapTrek (Experimental)
  Interventions: Behavioral: MapTrek

INTERVENTIONS:
Behavioral: MapTrek — Participants will receive a Fitbit activity monitor and access to the MapTrek game which will be visible on monitors set up in the residential facility.

SUMMARY:
Older adults are a growing population, with projections to reach 83.7 million by 2050. Furthermore, older adults are the most sedentary and least physically active adult population. It is estimated that nearly 90% of older adults 65 years of age or older do not meet the recommended levels of physical activity. Evidence suggests great health benefits can be achieved for older adults who are the most sedentary, and that replacing sitting with even light intensity walking can be beneficial.

The overarching goal of the project is to develop an inexpensive and scalable tool to increase volume of physical activity in our target population, older adults living in a residential facility. MapTrek is a web-based application that allows participants to take a virtual walk in interesting locations around the world while tracking their progress against the progress of other older adults living in a retirement community. Steps are counted using a commercially available accelerometer (e.g., Fitbit), and participants see their progress overlaid on Google Maps.

DETAILED DESCRIPTION:
All participants will be provided with a Fitbit activity monitor and instructed to wear it 24 hours/day (except for bathing/swimming time) on their wrist for 12 weeks. Participants will participate in four team-based walking races, each two weeks long. Participants will view their team progress on TV monitors placed in various locations at the Oaknoll facility. The Oaknoll leadership has given the research team approval to do this at their facility. The monitors will present aggregated team data and will not report any individual data that could link back to the individual participant.

At the end of the 8 week active intervention, research team members will meet with participants at Oaknoll to administer an exit/process evaluation survey. The exit survey will ask about psychosocial predictors of physical activity as well as participants thoughts and opinions of the MapTrek game. This survey should take approximate 10-15 minutes to complete. The participants will then be asked to wear the Fitbit for four more weeks without playing MapTrek, which will act as a control condition since this is a single-arm study.

The specific aims of the study are:

1. To determine the efficacy of MapTrek for improving physical activity levels of older adults living in a residential facility from baseline to 8 weeks.
2. To determine the efficacy of MapTrek for improving psychosocial outcomes(e.g., self-efficacy, social support, outcome expectations, social isolation) among older adults living in a residential facility from baseline to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, participants much be between 25 and 100 years of age, physically able to walk without limitations

Exclusion Criteria:

* Patients with cognitive or physical limitations that prohibit walking and visual or cognitive impairments causing inability to read.

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2019-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Carr, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from June 17, 2019 to June 27, 2019, by word of mouth and through advertisements posted on digital monitors located throughout the retirement community.
Pre-assignment Details: After providing their consent to participate, participants were asked to complete a baseline survey and provided a Fitbit activity monitor to wear for a minimum of 7 days to assess their baseline physical activity.
Groups:
- MapTrek: MapTrek: Participants will receive a Fitbit activity monitor and access to the MapTrek game for 8 weeks which will be visible on monitors set up in the residential facility.
Period: Overall Study
Arm/Group | MapTrek
Started | 68
Completed | 54
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | MapTrek
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 54
Age, Continuous [Mean (Full Range); unit: years] | 81.2 [68 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 54
Physical Activity [Mean (Inter-Quartile Range); unit: Steps/day] | 5438 [4620 to 6256]
Self-efficacy [Mean (Standard Deviation); unit: units on a scale] — cumulative score (0-90); higher=better
  units on a scale | 73.2 (14.1)
Social Support [Mean (Standard Deviation); unit: units on a scale] — mean score (0-4 range; higher = better)
  units on a scale | 2.2 (0.7)
Outcome Expectations [Mean (Standard Deviation); unit: units on a scale] — mean score (1-5 range) lower=better
  units on a scale | 4.4 (0.6)
Social Isolation [Mean (Standard Deviation); unit: units on a scale] — cumulative score (4-20) higher=better
  units on a scale | 17.9 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity
Description: Daily steps
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: Steps/day
Arm/Group | MapTrek
Number analyzed (Participants) | 54
Steps/day | 6681 [5840 to 7522]
Statistical Analysis 1: Comparison: MapTrek; In order to test the effect of the intervention on physical activity, linear mixed models examined changes in steps per day from study baseline (week 0) to the end of the active intervention (week 8); Test type: Superiority; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = .01

2. Secondary Outcome: Self-efficacy
Description: Self-efficacy was measured with the Self-Efficacy for Exercise scale, a 13-item questionnaire designed to assess participants' self-efficacy related to their ability to continue exercising in the face of barriers.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: cumulative score (0-90); higher=better
Arm/Group | MapTrek
Number analyzed (Participants) | 54
cumulative score (0-90); higher=better | 67.4 (15.2)

3. Secondary Outcome: Social Support
Description: Social support for physical activity was measured with a modified version of the Social Support and Exercise Survey. The Social Support and Exercise Survey is a 12-item (originally 13 item) questionnaire that assesses the level of support from family and friends that participants have in making health behavior changes (exercise)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mean score (0-4 range); higher=better
Arm/Group | MapTrek
Number analyzed (Participants) | 54
mean score (0-4 range); higher=better | 2.2 (0.8)

4. Secondary Outcome: Outcome Expectations
Description: Outcome expectations were measured with the Outcome Expectations for Exercise Scale. The Outcome Expectations for Exercise is a valid and reliable 9-item scale that assesses the participant's outcome expectations and benefits associated with exercise.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mean score (1-5 range) lower=better
Arm/Group | MapTrek
Number analyzed (Participants) | 54
mean score (1-5 range) lower=better | 4.4 (0.6)

5. Secondary Outcome: Social Isolation
Description: Social isolation was measured with a modified version of the Friendship Scale. The Friendship Scale is a 5-item (originally 6-item) scale that assesses 6 dimensions contributing to social isolation
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: cumulative score (4-20) higher=better
Arm/Group | MapTrek
Number analyzed (Participants) | 54
cumulative score (4-20) higher=better | 17.6 (2.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | MapTrek
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT04041869/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04041869/ICF_001.pdf